CLINICAL TRIAL: NCT04245163
Title: Development and Implementation of an Educational Program to Enhance Adherence to Glaucoma Treatment: A Mixed Method Study
Brief Title: Development and Implementation of an Educational Program to Enhance Adherence to Glaucoma Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Maria Achilleos, Principal investigator, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CUT15012018MA
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Glaucoma
Keywords: medication adherence; education*; intervention
MeSH Terms: conditions — Glaucoma; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants who will be randomized in control group will receive normal care (the care that each clinic provides to the patients) and will be given an educational material (without telling them that they are in the control group). They will receive, however, the education class later (at the end of the study). Participants in the intervention group will be invited for the training program
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will be invited for the training program.
  Interventions: Behavioral: Educational program
- Control Group (No Intervention): Participants who will be randomized in control group will receive normal care (the care that each clinic provides to the patients) and will be given an educational material (without telling them that they are in the control group). They will receive, however, the education class later (at the end of the study).

INTERVENTIONS:
Behavioral: Educational program — The intervention program will include 3 phases. At phase 1 a presentation on Microsoft PowerPoint in order to increase the general knowledge about glaucoma. At phase 2 a video and a one on one teaching to develop skills of administering the eye drops in a correct and systematic way. At phase 3, a discussion in order to identify cues to action that can easily be adopted by the patient in his/her daily routine, (such as, how to remember to put in drops) will take place.
  Arms: Intervention Group

SUMMARY:
This study evaluates the addition of an educational intervention program in order to improve medication adherence in glaucoma patients. Half of the participants will receive the educational program while the other half will receive normal care and a leaflet about glaucoma.

DETAILED DESCRIPTION:
Introduction. As the world population ages, glaucoma is becoming an increasingly significant cause of blindness. Statistics gathered by WHO in 2010, show that glaucoma is the leading cause of irreversible blindness, worldwide. A key component in the management of glaucoma, is the use of prescribed medications· but the effectiveness of medications depends on patient's adherence to treatment. However, there is evidence of poor adherence to prescribed medication in chronic diseases and a causative factor for that is the limited education and the low health literacy. This study aims to investigate the reasons of non-adherence to the medication plan among patients with glaucoma and secondly, according the findings, to develop and implement a comprehensive educational program.

Methods and analysis. This is a mixed method study which include 3 stages: a descriptive study (stage 1), focus group discussion (stage 2) and a randomised control trial (stage 3). Sample: Patients with glaucoma, using at least one kind of drops, will be recruited from the two ophthalmology clinics in Cyprus. Selected measures include: Glaucoma Treatment Compliance Assessment Tool (GTCAT), European Health Literacy Survey Questionnaire (HLS-EU-Q6) and the Glaucoma Medication Self-Efficacy Questionnaire (GMSEQ). The data will be analysed by SPSS program with descriptive and inferential statistics. Content analysis will be used for the data from the focus groups.

Ethics and dissemination. Permission to conduct the study received from the Cyprus National Bioethics Committee (ΕΕΒΚ ΕΠ 2019.01.220) and the board of management of the two ophthalmology clinics. All participants will be informed fully on the purpose and methods of the study. Consent forms will be signed and at any time participants will have the right to withdraw. Confidentiality of the participants will be respected as also the protection of data. Dissemination strategy includes presentations in international and national scientific conferences and publications in scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Ability to read and understand Greek
* Able to give informed consent
* Diagnosis of glaucoma or ocular hypertension, requiring treatment with hypotensive eye drops (at least one time per day).
* Patients who scored less than 80% adherent on GTCAT

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change to the Glaucoma Treatment Compliance Assessment Tool (GTCAT-28) | T0: before intervention (4-12 months before), T1: immediately after the intervention (same day), T2: One month after the intervention, T3: Three months after the intervention
  Easy and quick questionnaire specially designed for patients with glaucoma. It contains 27 statements with 5-interval Likert-type scale response (eg, 1- disagree a lot, 5-agree a lot) and 1 open ended question for assessing the knowledge, the Health Belief Model components (Barriers, Benefits, Cues to Action, Self-efficacy, Severity, Susceptibility), the patient-physician relationship, and their physical and mental health. The correct answers range from 0 to 27, with the highest score indicating more adherence to the treatment. The purpose is to assess the change between several time points (e.g. before the intervention, after the intervention-same day, one month after the intervention and three months after the intervention). The reason is, firstly, to assess if there is a change between T0 and T1 and secondly to assess if the effect of the intervention (as indicated by the change in the GTCAT) remain for a longer period of time.

SECONDARY OUTCOMES:
European Health Literacy Survey Questionnaire (HLS-EU-Q6) | T0: before the intervention (4-12 months before)
  The HLS-EU-Q6, includes 6 statements with 5-interval Likert-type scale response (eg, 1- disagree a lot, 5-agree a lot). We will use the HLS-EU-Q6 to assess the level of Health Literacy among the participants.
Change to the Glaucoma Medication Self-Efficacy Questionnaire (GMSEQ-16) | T0: before the intervention (4-12 months before), T1: immediately after the intervention (same day), T2: One month after the intervention, T3: Three months after the intervention
  The GMSEQ consists of 10 questions assessing Self-Efficacy in Glaucoma medication in general and 6 questions assessing Self-Efficacy in the eye drop technique. The response categories are: 'not at all confident', 'somewhat confident', 'very confident' and 'does not apply'. The purpose is to assess the change between several time points (e.g. before the intervention, after the intervention-same day, one month after the intervention and three months after the intervention). The reason is to assess firstly if there is a change (between T0 and T1) and secondly to asses if the effect of the intervention (as indicated by the change in the GMSEQ-16) remain for a longer period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Pantheon Eye Center, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No